CLINICAL TRIAL: NCT03134599
Title: Comparison of Clinical Performance and Subjective Preference Out of Three Cosmetic Contact Lenses (Limbal Ring-enhancing Lenses, LRE Lenses)
Brief Title: Comparison of Clinical Performance and Subjective Preference of Three Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CV_BSCHU
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Results first posted 2019-02-22 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- etafilcon A (Active Comparator)
  Interventions: Device: etafilcon A
- methafilcon A - Interozzo (Active Comparator)
  Interventions: Device: methafilcon A - Interozzo
- methafilcon A - CVI (Active Comparator)
  Interventions: Device: methafilcon A - CVI (CooperVision)

INTERVENTIONS:
Device: etafilcon A — contact lens
  Arms: etafilcon A
Device: methafilcon A - Interozzo — contact lens
  Arms: methafilcon A - Interozzo
Device: methafilcon A - CVI (CooperVision) — contact lens
  Arms: methafilcon A - CVI

SUMMARY:
The purpose of this study is to evaluate the clinical performance and subject's preference out of three LRE (Limbal Ring Enhancing) lens types: etafilcon A (Johnson&Johnson), methafilcon A (Interozzo), and methafilcon A (CooperVision).

DETAILED DESCRIPTION:
This will be a subject-masked, bilateral, randomized, crossover dispensing study to compare clinical performance and subjective preference out of three lens types. Sixty subjects will be assigned into three groups and each group will wear the test and control lenses as matched pairs for one week in random order. Lenses will be worn on a daily wear, daily disposable schedule.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and above and has full legal capacity as a volunteer Understand the rights as a research subject and willing and able sign a statement of informed consent
* Existing soft contact lens wearers or previous experience of contact lens wear
* Being able to wear the study lenses for at least eight hours a day
* At least 6/9 visual acuity in each eye with the study lenses
* Astigmatism less than 1.50 D (Diopter) in both eyes
* Agreed to follow the protocol and not to participate in other clinical research for the duration of this study

Exclusion Criteria:

* Have an ocular disorder which would normally contraindicate contact lens wear
* Have a systemic disorder or any infectious diseases which would normally contraindicate contact lens wear
* Have previously had any ocular surgery such as corneal refractive surgery
* Have less than 6/9 visual acuity in each eye with the study lenses
* Are currently using any topical medication such as eye drops or ointment
* Have any corneal distortion resulting from previous rigid lens wear or have keratoconus
* Are currently pregnant or lactating
* No previous contact lens wear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-06-24 (Actual); Study Completion 2017-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Optometry & Vision Science, Catholic University of Daegu, Korea (Rep), Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Etafilcon A, Methafilcon A-Interozzo, Methafilcon A (CVI): etafilcon A first, then methafilcon A - Interozzo then methafilcon A (CVI) contact lens
- Etafilcon A, Methafilcon A (CVI), Methafilcon A-Interozzo: etafilcon A first, then methafilcon A (CVI) then methafilcon A - Interozzo contact lens
- Methafilcon A-Interozzo, Methafilcon A (CVI), Etafilcon A: methafilcon A - Interozzo first, then methafilcon A (CVI), then etafilcon A contact lens
- Methafilcon A-Interozzo, Etafilcon A Methafilcon A (CVI): methafilcon A - Interozzo first, then etafilcon A contact lens, then methafilcon A (CVI)
- Methafilcon A (CVI), Methafilcon A-Interozzo, Etafilcon A: methafilcon A (CVI) first, then methafilcon A - Interozzo, then etafilcon A contact lens
- Methafilcon A (CVI), Etafilcon A, Methafilcon A-Interozzo: methafilcon A (CVI) first, then etafilcon A contact lens, then methafilcon A - Interozzo
Period: Week 1
Arm/Group | Etafilcon A, Methafilcon A-Interozzo, Methafilcon A (CVI) | Etafilcon A, Methafilcon A (CVI), Methafilcon A-Interozzo | Methafilcon A-Interozzo, Methafilcon A (CVI), Etafilcon A | Methafilcon A-Interozzo, Etafilcon A Methafilcon A (CVI) | Methafilcon A (CVI), Methafilcon A-Interozzo, Etafilcon A | Methafilcon A (CVI), Etafilcon A, Methafilcon A-Interozzo
Started | 10 | 10 | 10 | 11 | 10 | 9
Completed | 10 | 10 | 10 | 11 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Period: Week 2
Arm/Group | Etafilcon A, Methafilcon A-Interozzo, Methafilcon A (CVI) | Etafilcon A, Methafilcon A (CVI), Methafilcon A-Interozzo | Methafilcon A-Interozzo, Methafilcon A (CVI), Etafilcon A | Methafilcon A-Interozzo, Etafilcon A Methafilcon A (CVI) | Methafilcon A (CVI), Methafilcon A-Interozzo, Etafilcon A | Methafilcon A (CVI), Etafilcon A, Methafilcon A-Interozzo
Started | 10 | 10 | 10 | 11 | 9 | 9
Completed | 9 | 10 | 10 | 10 | 8 | 9
Not Completed | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 1 | 0
Period: Week 3
Arm/Group | Etafilcon A, Methafilcon A-Interozzo, Methafilcon A (CVI) | Etafilcon A, Methafilcon A (CVI), Methafilcon A-Interozzo | Methafilcon A-Interozzo, Methafilcon A (CVI), Etafilcon A | Methafilcon A-Interozzo, Etafilcon A Methafilcon A (CVI) | Methafilcon A (CVI), Methafilcon A-Interozzo, Etafilcon A | Methafilcon A (CVI), Etafilcon A, Methafilcon A-Interozzo
Started | 9 | 10 | 10 | 10 | 8 | 9
Completed | 9 | 10 | 10 | 9 | 8 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants wore enfilcon A, methafilcon A (Interozzo) and methafilcon A (CooperVision) contact lenses.
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 60

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Subjective ratings of comfort for each lens pair was assessed. Scale 0-100, 0=causes pain, 100=very comfortable.
Time Frame: 1 week per intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Etafilcon A: etafilcon A contact lens
Arm/Group | Etafilcon A | Methafilcon A - Interozzo | Methafilcon A - CVI
Number analyzed (Participants) | 54 | 54 | 54
units on a scale | 64.19 (21.70) | 58.57 (22.48) | 59.31 (21.53)

ADVERSE EVENTS:
Time Frame: 1 week per intervention, 3 weeks total
Groups:
- Etafilcon A: All subjects who wore etafilcon A contact lenses as either the first, second or third pair.
- Methafilcon A-Interozzo: All subjects who wore methafilcon A-Interozzo contact lenses as either the first, second or third pair.
- Methafilcon A (CVI): All subjects who wore methafilcon A (CVI) contact lenses as either the first, second or third pair.
Arm/Group | Etafilcon A | Methafilcon A-Interozzo | Methafilcon A (CVI)
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the sponsor should be notified of any results communications and has ability to review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03134599/Prot_SAP_001.pdf